CLINICAL TRIAL: NCT01444989
Title: Development and Validation of a Quality of Life Instrument for Actinic Keratosis
Acronym: AKRQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00017619
Record Dates: First submitted 2011-09-29; First posted 2011-10-03 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Actinic Keratosis
Keywords: "Sun spots"; "Pre-cancerous skin lesion"
MeSH Terms: conditions — Keratosis, Actinic; Melanosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients without actinic keratosis (Experimental): Patients with out the diagnosis of actinic keratosis will receive the experimental questionnaire.
  Interventions: Other: AKRQ questionnaire; Other: Skindex-16, DLQI, Skin Health Calculator
- Patients with Actinic Keratosis (Experimental): Patients with the diagnosis of actinic keratosis will receive the experimental questionnaire.
  Interventions: Other: AKRQ questionnaire; Other: Skindex-16, DLQI, Skin Health Calculator

INTERVENTIONS:
Other: AKRQ questionnaire — The AKRQ is an experimental instrument composed of 10 questions that assess quality of life and risk factors
Other: Skindex-16, DLQI, Skin Health Calculator — These are all previously validated questionnaires

SUMMARY:
Actinic keratoses (AKs) are some of the most common lesions seen by dermatologists. Flesh colored to erythematous, these lesions often present with scaling or crusting in sun damaged regions of the body. While they are physically visible and often palpable, these changes can also result in psychosocial changes in patients, including embarrassment about their skin or reduction in leisure activities to avoid further sun exposure. At the same time, AKs are known to progress in a significant number of cases to squamous cell carcinoma (SCC), a concern in terms of its metastatic potential.

The primary purpose of developing this questionnaire is to examine how well it can potentially identify patients with actinic keratoses. However, since AK is associated with significant detriment to quality of life for validity/reliability assessment, the investigators propose to give a compilation of four self-assessment questionnaires (not specific to AK but validated for skin health in general) to subjects with at least one actinic keratosis and age- and sex- matched participants without AKs, defined as the control population. These will include the SKINDEX-16, the DLQI and the Skin Health Calculator, as well as a questionnaire composed of items specific to predisposition to AKs to be able to better assess the discriminatory power of the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or older being seen in a dermatology clinic
* Informed consent of participation must be given by subject

Exclusion Criteria:

* Inability to complete all study questionnaires.
* Subjects who are unable to read and write English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Difference in questionnaire score in patients with Actinic keratosis and with out actinic keratosis | Baseline
  We are developing an actinic keratosis risk assessment questionnaire and is designed to distinguish patients who have a higher likelihood of having a diagnosis of actinic keratosis. The outcome measure is the difference in scores between those with actinic keratosis and those without.

SECONDARY OUTCOMES:
Correlation between AKRQ and DLQI scores | Baseline
  The DLQI is a validated instrument. We will report how well our new instrument correlates with the DLQI.
The correlation between AKRQ and Skindex-16 scores | Baseline
  The Skindex-16 is a validated instrument. We will report how well our new instrument correlates with the Skindex-16.
The correlation between the AKRQ and Skin Health Calculator scores. | Baseline
  The Skin health calculator is a validated instrument. We will report how well our new instrument correlates with the Skin Health Calculator

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Health Sciences Dermatology, Winston-Salem, North Carolina, United States